CLINICAL TRIAL: NCT06413498
Title: A Phase 3, Randomized, Open-Label Study to Compare the Efficacy and Safety of Anitocabtagene Autoleucel Versus Standard of Care Therapy in Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study Comparing Anitocabtagene Autoleucel to Standard of Care Therapy in Participants With Relapsed/ Refractory Multiple Myeloma
Acronym: iMMagine-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Collaborators: Arcellx, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-679-0788; 2024-511188-26 (Other: European Medicines Agency); jRCT2043240170 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; CAR-T; ddBCMA; BCMA
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; pomalidomide; Bortezomib; Dexamethasone; daratumumab; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anitocabtagene Autoleucel (Experimental): Participants with RRMM will receive lymphodepletion chemotherapy with cyclophosphamide and fludarabine for 3 days followed by single dose of anitocabtagene autoleucel chimeric antigen receptor positive (CAR+) on Day 1.
  Interventions: Drug: Anitocabtagene Autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Standard of Care Therapy (SOCT) (Active Comparator): Participants will receive the investigator's choice of one of the following therapies:
  * pomalidomide, bortezomib, and dexamethasone (PVd) (21-day cycles)
  * daratumumab, pomalidomide, and dexamethasone (DPd) (28-day cycles)
  * carfilzomib, daratumumab, and dexamethasone (KDd) (28-day cycles)
  * carfilzomib and dexamethasone (Kd) (28-day cycles)
  Interventions: Drug: Pomalidomide; Drug: Bortezomib; Drug: Dexamethasone; Drug: Daratumumab; Drug: Carfilzomib

INTERVENTIONS:
Drug: Anitocabtagene Autoleucel — A single infusion of CAR+ transduced autologous T cells
  Other Names: CART-ddBCMA
  Arms: Anitocabtagene Autoleucel
Drug: Cyclophosphamide — Administered intravenously
  Arms: Anitocabtagene Autoleucel
Drug: Fludarabine — Administered intravenously
  Arms: Anitocabtagene Autoleucel
Drug: Pomalidomide — Tablet administered orally
  Arms: Standard of Care Therapy (SOCT)
Drug: Bortezomib — Administered intravenously or subcutaneously
  Arms: Standard of Care Therapy (SOCT)
Drug: Dexamethasone — Tablet administered orally
  Arms: Standard of Care Therapy (SOCT)
Drug: Daratumumab — Administered intravenously or subcutaneously
  Arms: Standard of Care Therapy (SOCT)
Drug: Carfilzomib — Administered intravenously
  Arms: Standard of Care Therapy (SOCT)

SUMMARY:
The goal of this study (iMMagine-3) is to compare the study drug, anitocabtagene autoleucel to standard of care therapy (SOCT) in participants with relapsed/refractory multiple myeloma who have received 1 to 3 prior lines of therapy, including an anti-CD38 monoclonal antibody and an immunomodulatory drug.

The primary objective of this study is to compare the efficacy of anitocabtagene autoleucel versus SOCT in participants with RRMM.

DETAILED DESCRIPTION:
After completing the treatment period, all participants who will receive anitocabtagene autoleucel, will be followed in the post-treatment follow-up period. Thereafter, participants will transition to a separate long-term follow-up study (KT-US-982-5968) to continue follow-up out to 15 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented historical diagnosis of multiple myeloma (MM)
* Received 1 to 3 prior lines of antimyeloma therapy, including an immunomodulatory drug (IMiD) and an anti-cluster of differentiation 38 (CD38) monoclonal antibody (mAb). A minimum of 2 consecutive cycles of an IMiD and an anti-CD38 mAb in any prior line of therapy is required. The IMiD and anti-CD38 mAb do not need to be from the same regimen in the prior line(s) of therapy.
* Documented evidence of progressive disease by IMWG criteria based on the investigator's determination on or within 12 months of the last dose of the last regimen
* Measurable disease at screening per IMWG, defined as any of the following:

  * Serum M-protein level ≥ 0.5 g/dL or urine M-protein level ≥ 200 mg/24 hours; or
  * Light chain MM without measurable disease in the serum or urine: serum free light chain ≥ 10 mg/dL and abnormal serum free light chain ratio
* Only individuals who are candidates to receive at least 1 of the 4 SOCT regimens (PVd, DPd, KDd, or Kd), as determined by the investigator, should be considered for this study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Females of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)

Key Exclusion Criteria:

* Prior B-cell maturation antigen (BCMA)-targeted therapy
* Prior T-cell engager therapy
* Prior CAR therapy or other genetically modified T-cell therapy
* Active or prior history of central nervous system (CNS) or meningeal involvement of MM
* Cardiac atrial or cardiac ventricular MM involvement
* History of or active plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or amyloidosis
* Active malignancy (other than MM) requiring ongoing treatment for disease control within the last 24 months. Myelodysplastic syndrome (even without ongoing treatment) is not permitted.
* Prior auto-SCT within 12 weeks before randomization
* Prior allogeneic stem cell transplant (allo-SCT)
* High-dose (eg, cumulative > 70 mg prednisone or equivalent) systemic steroid therapy or any other form of immunosuppressive therapy within 14 days before randomization
* Live vaccine ≤ 4 weeks before randomization
* Contraindication to fludarabine or cyclophosphamide
* History of allergy or hypersensitivity to any study agent or study drug components. Individuals with a history of severe hypersensitivity reaction to dimethyl sulfoxide (DMSO) are excluded.
* Life expectancy < 12 weeks

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 4 years
  PFS is defined as the time from randomization to disease progression per International Myeloma Working Group (IMWG) criteria as determined by independent review committee (IRC), or death due to any cause, whichever occurs first.
Minimal Residual Disease (MRD) Complete Response (CR) Rate at 9 Months | Up to 9 months
  Minimal MRD is defined as the proportion of participants achieving CR/stringent CR (sCR) and MRD-negative status at 9 months. MRD negativity at 9 months is defined as negative MRD value at 9 months (± 3 months) in bone marrow assessment (< 1 in 105 nucleated cells per IMWG criteria using NGS) (Kumar 2016). CR/sCR per IMWG criteria is determined by IRC.

SECONDARY OUTCOMES:
CR Rate (CR/ Stringent Complete Response (sCR)) | Up to 4 years
  CR rate is defined as the proportion of participants who achieved a best overall response of CR or sCR per IMWG criteria as determined by IRC.
Overall MRD Negativity | Up to 7 years
  Overall MRD negativity, defined as the proportion of any MRD negativity in participants with bone marrow aspirate (< 1 in 10^5 nucleated cells per IMWG criteria using next-generation sequencing (NGS)) at any time after randomization until disease progression, subsequent anti-multiple myeloma (MM) therapy, or death.
Overall survival (OS) | Up to 7 years
  OS is defined as the time from randomization to death due to any cause.
Overall Response Rate (ORR) | Up to 7 years
  ORR is defined as the proportion of participants who achieve a best overall response of at least partial response (PR) or better (sCR, CR, very good partial response (VGPR), or PR) per IMWG criteria.
MRD-negative CR/sCR | Up to 7 years
  MRD-negative CR/sCR is defined as the proportion of participants achieving MRD-negative CR/sCR until disease progression, subsequent anti-MM therapy, or death.
MRD-negative VGPR+ | Up to 7 years
  MRD-negative VGPR+ is defined as the proportion of participants achieving MRD negativity and sCR/CR/VGPR until disease progression, subsequent anti-MM therapy, or death.
Sustained MRD Negativity | Up to 7 years
  Sustained MRD negativity is defined as the proportion of participants remaining MRD-negative at the 10^-5 sensitivity threshold for the specified number of months starting from the first MRD-negative assessment date to the last MRD-negative assessment date prior to disease progression, subsequent anti-MM therapy, or death. Duration may include ≥ 12 months. Sustained MRD negativity will be evaluated for overall MRD negativity, MRD-negative CR/sCR, and MRD-negative VGPR+.
Duration of Response (DOR) | Up to 7 years
  DOR is derived only among participants who experience an overall response (sCR, CR, VGPR, or PR) per IMWG criteria and is defined as the time from first overall response to disease progression per IMWG criteria, or death from any cause, whichever occurs first.
Time to Progression | Up to 7 years
  Time to progression is defined as the time from randomization to the first documented disease progression per IMWG criteria, or death due to disease progression, whichever occurs first.
Time to Next Treatment | Up to 7 years
  Time to next treatment is defined as the time from randomization to the start of subsequent anti-MM therapy or death from any cause, whichever occurs first.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose up to 7 years
Percentage of Participants With Anti-Anitocabtagene Autoleucel CAR Antibodies (Anitocabtagene Autoleucel Arm) | Up to 7 years
Percentage of Participants With Presence of Replication-Competent Lentivirus (Anitocabtagene Autoleucel Arm) | Up to 7 years
Change From Baseline in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | Up to 7 years
  The EORTC-QLQ-C30 is a multi-item questionnaire measuring the following content: five (5) multi-item functional scales, three (3) multi-item symptom scales, six (6) single item symptoms scales, one (1) global health status scale, and one (1) global health-related quality of life (HRQoL). Each scale is measured from 0 to 100 after a linear transformation. Higher scores for functioning scales and for the Global Health Status or Global HRQoL scales indicate a higher level of functioning and a better HRQoL respectively, whereas higher scores in symptom scales represent a high level of symptoms.
Change From Baseline in the EORTC - Multiple Myeloma Module (EORTC QLQ-MY20) Score | Up to 7 years
  The EORTC QLQ-MY20 has 20 items across 4 independent subscales; 2 functional subscales (body image, future perspective), and 2 symptoms scales (disease symptoms, and side effects of treatment) with a recall period of one week. Scores from each subscale are transformed from 0 to 100. For the functional scales, high scores represent improvement. For the symptom scales, higher scores represent worsening.
Change From Baseline in the European Quality of Life 5-Dimension 5-Level Scale (EQ-5D-5L) Score | Up to 7 years
  The EQ-5D-5L questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L comprises 2 components: a questionnaire covering 5 dimensions and a tariff of values based upon direct valuations of health states using a visual analog scale (VAS). The total score for EQ-5D-5L index is presented on a range where higher scores indicate better outcome. A positive change from Baseline indicates improvement.
Percentage of Participants Using Healthcare Resources | Up to 7 years
  Healthcare resource utilization will be assessed based on the numbers of hospitalizations, intensive care unit (ICU) inpatient days, and non-ICU inpatient days.

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (119):
- United States (47):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital, Gilbert, Arizona
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Moores Cancer Center, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - UCLA Hematology/Oncology (Bowyer Infusion Clinic), Santa Monica, California
  - Stanford Cancer Institute, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Sylvester Comprehensive Cancer Center, Coral Gables, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Southeastern Regional Medical Center, Inc. dba City of Hope Atlanta, Newnan, Georgia
  - St. Luke's Cancer Institute, Boise, Idaho
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - IU Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Corewell Health - Lemmen-Holton Cancer Pavilion, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists - Legacy, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New Mexico Cancer Research Alliance, Albuquerque, New Mexico
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Weill Cornell Medicine - New York Presbyterian Hosptial, New York, New York
  - Novant Health Cancer Institute - Hematology, Charlotte, North Carolina
  - Novant Health Cancer Institute Hematology- Forsyth, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Tennessee Oncology, PLLC - Greco-Hainsworth Centers for Research, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Houston Methodist Hospital Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Epworth HealthCare, Richmond, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (4):
  - Ordensklinikum Linz GmbH Elisabethinen, Hamatologie mit Stammzelltransplantation, Hamostaseologie und medizinische Onkologie, Linz
  - Paracelsus Medizinischen Privatuniversitaet, Salzburg
  - University Hospital St. Poelten, Department of Internal Medicine I, Sankt Pölten
  - Medical University of Vienna, Vienna
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital of Antwerp, Edegem
  - UZ Leuven, Flemish Brabant
  - UZ Gent, Gent Oost-Vlaanderen
- Canada (4):
  - QEII Health Sciences Centre, Halifax
  - McGill University Health Center, Montreal
  - The Ottawa Hospital - General Campus, Ottawa
  - University Health Network - The Princess Margaret Cancer Centre, Toronto
- Fakultni Nemocnice Ostrava, Severomoravsky KRAJ, Czechia
- France (10):
  - CHU de Lille- Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU De Montpellier - Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de Toulouse. IUCT Oncopole, Toulouse
- Germany (7):
  - Universitatsklinikum Koln, Klinik I fOr lnnere Medizin, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Universitatsklinikum Leipzig, Leipzig
  - TUM Klinikum, Rechts der Isar, Klinik und Poliklinik fur Innere Medizin III, Hamatologie und Onkologie, München
  - Universitatsklinikum Wurzburg, Tübingen
- Italy (5):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - IRCCS AOU di Bologna, Bologna
  - Ospedale San Raffaele, Milan
  - Policlinico Universitario Argostino Gemelli, Roma
  - AOU Città della Salute e della Scienza Presidio Ospedaliero Molinette, Torino
- Japan (7):
  - Hyogo Medical University Hospital, Hyōgo
  - Nagoya City University Hospital, Nagoya
  - The University of Osaka Hospital, Osaka
  - Hamamatsu University Hospital, Shizuoka
  - Jichi Medical University Hospital, Tochigi
  - Juntendo University School of Medicine Juntendo Clinic, Tokyo
  - Japanese Red Cross Medical Center, Tokyo
- Netherlands (3):
  - Amsterdam UMC - Location vUmc, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- Poland (3):
  - Warszawa-Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw
- Spain (11):
  - ICO Badalona-H.U. Germans Trias i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Switzerland (2):
  - Inselspital - Universitätsspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- United Kingdom (6):
  - University Hospitals Bristol NHS Foundation Trust, Bristol Haematology and Oncology Centre, Bristol
  - University Hospital of Wales, Cardiff
  - Leeds Teaching Hospitals NHS Trust, St James's University Hospital, Leeds
  - King's College Hospital, London
  - University College London Hospital, London
  - Newcastle Hospitals NHS Foundation Trust, Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06413498